CLINICAL TRIAL: NCT05003336
Title: Effects of Xiangshao Granules on Anxiety in Menopausal Women: A Multicenter, Randomized, Double-blind, Placebo-controlled Study.
Brief Title: Effects of Xiangshao Granules on Anxiety in Menopausal Women.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XSKL20200422
Record Dates: First submitted 2021-08-10; First posted 2021-08-12 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-08

CONDITIONS: Anxiety; Menopause
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xiangshao Granules (Experimental): dissolve 1 sachet (4 g) of Xiangshao Granules in water to be drank 3 times a day after meal for 8 weeks
  Interventions: Drug: Xiangshao Granules
- Xiangshao Granules Placebo (Placebo Comparator): dissolve 1 sachet (4 g) of Xiangshao Granules placebo in water to be drank 3 times a day after meal for 8 weeks
  Interventions: Drug: Xiangshao Granules Placebo

INTERVENTIONS:
Drug: Xiangshao Granules — dissolve 1 sachet (4 g) in water to be drank 3 times a day after meal for 8 weeks
  Arms: Xiangshao Granules
Drug: Xiangshao Granules Placebo — Xiangshao Granules Placebo
  Arms: Xiangshao Granules Placebo

SUMMARY:
Symptoms of anxiety are prevalent during the menopausal transition and early postmenopause. These symptoms are mainly improved by anti-anxiety agents, which are associated with some adverse effects including dizziness, sleepiness, and constipation and not all patients respond to currently available pharmacological treatments, thus novel agents with fewer side effects are needed. Some studies have shown that traditional Chinese medicine can alleviate menopausal symptoms safely and economically, and improve quality of life. Xiangshao granules reportedly have good curative effects on menopausal symptoms and premenstrual syndrome and exhibit good safety. This study aim to evaluate the efficacy and safety of Xiangshao granule in improving anxiety state of women with menopause syndrome.

ELIGIBILITY:
Inclusion Criteria:

* meet the diagnostic criteria for menopause syndrome (age 40-65 years, being in the menopausal transition stage or postmenopausal stage determined according to the 2011 Stages of Reproductive Aging Workshop +10 criteria).
* 50 ≤ SAS scores ≤ 69.
* improved Kupperman scores ≥16.
* has an intact uterus and at least one ovary.
* able and willing to participate in study and provide written informed consent, and agrees to follow all study requirements. The investigator consider the subject able to complete the study.

Exclusion Criteria:

* history of allergy or sensitivity to investigational product.
* currently or historically taking medication or psychotherapy for menopause anxiety in the past 4 weeks, including but not limited to estrogens, oestrogen-like hormone, Chinese medicine or health care products used to relieve anxiety (such as soy isoflavones, vitamin E, black cohosh), anti-anxiety agents, antidepressants, mood stabilizers, sedatives.
* anxiety or other psychiatric disease unrelated to menopause (eg., currently or previously diagnosed as major depression, acute panic disorder, obsessive-compulsive disorder, phobia, hypochondria, mood disorder or schizophrenia or psychiatric diseases caused by other psychoactive substances or organic diseases), anxiety symptoms caused by stress, suicidal tendency, alcohol or drug dependence, etc.
* having major depression as defined by a SDS score≥70 at screening.
* systemic disease (eg., hypothyroidism/hyperthyroidism, unstable coronary heart disease, severe hypertension [sbp≥180mmHg and/or dbp≥110mmHg] or pheochromocytoma).
* definite diagnosis of endometrial cancer, cervical cancer, ovarian cancer and other gynecological malignancies, as well as breast cancer.
* severe liver or kidney diseases (eg., alanine aminotransferase[ALT]/aspartate aminotransferase[AST]/serum creatinine[Scr] levels 2 times greater than the upper limit of normal) or severe primary diseases in cardiovascular, cerebrovascular, liver, kidney and hematopoietic system.
* participated in other clinical trials within the last 3 months.
* lactating or pregnant women, or plan to become pregnant during study or not agree to use reliable contraceptive methods throughout the study period.
* other reasons the investigator consider the patient may not be suitable for the study.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2021-12-23 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Self-rating Anxiety Scale (SAS) scores change (%) | 8 weeks
  % change in SAS scores after 8 weeks of treatment compared with baseline scores

SECONDARY OUTCOMES:
SAS scores change (%) | 4 weeks
  % change in SAS scores after 4 weeks of treatment compared with baseline scores
Kupperman scores change (%) | 4 weeks
  % change in Kupperman scores after 4 weeks of treatment compared with baseline scores
Kupperman scores change (%) | 8 weeks
  % change in Kupperman scores after 8 weeks of treatment compared with baseline scores
Self-rating Depression Scale (SDS) scores change (%) | 4 weeks
  % change in SDS scores after 4 weeks of treatment compared with baseline scores
SDS scores change (%) | 8 weeks
  % change in SDS scores after 8 weeks of treatment compared with baseline scores
serum Follicle Stimulating Hormone (FSH) level | 4 weeks
  change in serum FSH level after 4 weeks of treatment compared with baseline
serum FSH level | 8 weeks
  change in serum FSH level after 8 weeks of treatment compared with baseline
serum estradiol (E2) level | 4 weeks
  change in serum estradiol(E2) level after 4 weeks of treatment compared with baseline
serum estradiol (E2) level | 8 weeks
  change in serum estradiol(E2) level after 8 weeks of treatment compared with baseline
gastrointestinal symptom score (GIS) change (%) | 4 weeks
  % change in GIS after 4 weeks of treatment compared with baseline scores
gastrointestinal symptom score (GIS) change (%) | 8 weeks
  % change in GIS after 8 weeks of treatment compared with baseline scores

CONTACTS AND LOCATIONS:
Overall Officials: Rong Chen, Principal Investigator — Peking Union Medical College Hospital
Locations (18):
- China (18):
  - Anhui Province Maternity & Child Health Hospital, Hefei, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Chongqing Health Center for Women and Children, Chongqing, Chongqing Municipality
  - Gansu Provincial Maternity and Child-care Hospital, Lanzhou, Gansu
  - Cangzhou People's Hospital, Cangzhou, Hebei
  - Second Hospital of Hebei Medical University, Shijiangzhuang, Hebei
  - The First Affiliated Hospital of Henan University, Kaifeng, Henan
  - Zhengzhou Central Hospital Affiliated to Zhengzhou University, Zhengzhou, Henan
  - Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Province Hospital of Chinese Medicine, Nanjing, Jiangsu
  - Taizhou People's Hospital, Taizhou, Jiangsu
  - Zhangjiagang First People's Hospital, Zhangjiagang, Jiangsu
  - Jiangxi Maternal and Child Health Hospital, Nanchang, Jiangxi
  - Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
  - School of Clinical medicine & The First Affiliated Hospital of Chengdu Medical College, Chengdu, Sichuan
  - Tianjin Hospital of ITCWM Nankai Hospital, Tianjin, Tianjin Municipality